CLINICAL TRIAL: NCT00444964
Title: Growth Hormone Use in Adults With Prader-Willi Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 303-C02R
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Primary Cohort (Experimental): Nutropin AQ
  Interventions: Drug: Nutropin AQ

INTERVENTIONS:
Drug: Nutropin AQ — 0.0125 mg/kg/day
  Other Names: Growth Hormone

SUMMARY:
The main research question this protocol aims to answer is whether treatment with growth hormone will impact body composition, quality of life, and energy balance in PWS adults, and if there is a loss of effects after cessation of treatment for at least 12 months.

DETAILED DESCRIPTION:
The main research question this protocol aims to answer is whether treatment with growth hormone will impact body composition, quality of life, and energy balance in PWS adults, and if there is a loss of effects after cessation of treatment for at least 12 months. Specific outcomes to be evaluated are as follows:

• Increased IGF-1 as a function of human growth hormone dosage compared with baseline.

1. Improvement of indicators or risk factors for co-morbid diseases [diabetes (by measuring insulin and glucose levels), cardiovascular disease (by measuring lipids and fatty acids), and pulmonary function] in participants.
2. Improvement in quality of life measures as indicated by ratings on established behavior checklists in participants.
3. Changes in body composition (decreased fat, increased lean body mass and bone density) as determined by DEXA in participants.
4. Increased energy expenditure as determined by whole-room calorimeter measures (8 hour energy expenditure, RMR, TEF, mechanical work); diet records, physical activity monitors and strength measures.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 60 years old
* Male or female with diagnosed Prader-Willi syndrome confirmed by genetic testing (e.g., mPCR)
* Low IGF-1 level (e.g.,≤25%) at baseline
* Ability to provide informed consent or availability of a suitable legally authorized representative

Exclusion Criteria:

* Pregnancy
* Previous treatment with growth hormone
* Uncontrolled endocrine disease, (i.e. diabetes or thyroid)
* History of severe scoliosis
* Heart disease
* Uncontrolled high blood pressure or history of stroke
* Morbid obesity (using PWS growth charts)
* Severe sleep apnea or known breathing difficulties/obstruction (as per history or diagnostic testing results

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2012-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merlin G Butler, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- The Children's Mercy Hospital, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Cohort
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Primary Cohort
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Body Composition
Description: Anthropometric Measures and Body Composition
Time Frame: 12 and 24 months
Population: All patients enrolled
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Primary Cohort
Number analyzed (Participants) | 11
percentage of body fat
  Baseline | 51.2 (2.1)
  12 Months | 48.5 (2.2)
  24 Months | 52.1 (2.3)
Statistical Analysis 1: Comparison: Primary Cohort; Test type: Other; p < 0.05, Mixed Models Analysis

2. Primary Outcome: Blood Chemistry
Description: Insulin-like growth factor I- IGF-1
Time Frame: 12 and 24 months
Population: All patients enrolled
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Primary Cohort
Number analyzed (Participants) | 11
ng/ml
  Baseline | 93 (37.6)
  12 months | 385 (48.6)
  24 Months | 140 (53.1)
Statistical Analysis 1: Comparison: Primary Cohort; Test type: Other; p < 0.05, Mixed Models Analysis

3. Primary Outcome: Physical Activity
Description: Duration of daily physical activity
Time Frame: 12 and 24 months
Population: All patients enrolled
Measure: Mean (Standard Deviation); unit: Minutes per Day
Arm/Group | Primary Cohort
Number analyzed (Participants) | 11
Minutes per Day
  Baseline | 177 (27)
  12 Months | 256 (33)
  24 Months | 215 (49)
Statistical Analysis 1: Comparison: Primary Cohort; Test type: Other; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Primary Cohort
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Cohort (N=11)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) — participant slipped in bowling alley and fractured tibia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes